CLINICAL TRIAL: NCT02237651
Title: Topical Nasopharyngeal Anesthesia in Outpatient Bronchoscopy
Brief Title: Topical Anesthesia / Bronchoscopy
Acronym: TNA
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: MHH 09/03/2014
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-04

CONDITIONS: Equally of Delivery Systems of Local Anesthesia in Bronchoscopy
Keywords: anesthesia; bronchosocopy; lung transplantation
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- topical anesthesia multi-use device: anesthesia with multi-use device (Laryngeal atomizer, Karl Storz, Tuttlingen, Germany
  Interventions: Device: topical anesthesia multi-use device
- topical anesthesia Intranasal Mucosal Atomization: single-use product (LMA® MAD Nasal™ Intranasal Mucosal Atomization Device, Teleflex medical, Kernen Germany) for topical anesthesia
  Interventions: Device: topical anesthesia Intranasal Mucosal Atomization

INTERVENTIONS:
Device: topical anesthesia multi-use device
  Other Names: anesthesia with multi-use device (Laryngeal atomizer, Karl Storz, Tuttlingen, Germany
  Groups: topical anesthesia multi-use device
Device: topical anesthesia Intranasal Mucosal Atomization
  Other Names: single-use product (LMA® MAD Nasal™ Intranasal Mucosal Atomization Device, Teleflex medical, Kernen Germany) for topical anesthesia
  Groups: topical anesthesia Intranasal Mucosal Atomization

SUMMARY:
The primary aim of this study is to compare a simplified single-use product (LMA® MAD Nasal™ Intranasal Mucosal Atomization Device, Teleflex medical, Kernen Germany) for topical nasopharyngeal anesthesia in comparison to a multi-use device (Laryngeal atomizer, Karl Storz, Tuttlingen, Germany in terms of patient self-rated nasopharyngeal symptoms.

DETAILED DESCRIPTION:
Patients included in the first half of the study (topical anesthesia with the Laryngeal atomizer) and with need for another bronchoscopy in the second half of the study (topical anesthesia with the Intranasal Mucosal Atomization Device) will be asked to repeat the questionnaire after the second bronchoscopy to allow in-patient comparison.

Description of the primary efficacy analysis and population:

The primary endpoint of patient self-rated anesthesia by visual analogue scale after topical nasopharyngeal anesthesia for bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients after lung transplantation (single, double or combined)
* Informed consent
* outpatient bronchoscopy

Exclusion Criteria:

* Oxygen requirement at rest
* Need for peri-interventional sedation
* limited German language skills or other reasons which might impair patient communication or computer handling

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Equally | 30 min.
  The primary endpoint of patient self-rated anesthesia by visual analogue scale after topical nasopharyngeal anesthesia for bronchoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fuehner, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Dep. Respiratory Medicine, Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Fuehner T, Fuge J, Jungen M, Buck A, Suhling H, Welte T, Gottlieb J, Greer M. Topical Nasal Anesthesia in Flexible Bronchoscopy--A Cross-Over Comparison between Two Devices. PLoS One. 2016 Mar 15;11(3):e0150905. doi: 10.1371/journal.pone.0150905. eCollection 2016. PMID 26978775